CLINICAL TRIAL: NCT02065167
Title: Evaluation of Safety and Feasibility of Bone Marrow Derived Autologous MSCs to Enhance Bone Healing in Patients With Avascular Necrosis of the Femoral Head
Brief Title: Evaluation of Mesenchymal Stem Cells to Treat Avascular Necrosis of the Hip
Acronym: ORTHO-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Prof Enrique Gomez-Barrena, Full Professor and Chair of orthopaedic surgery, Universidad Autonoma de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO -2; 2012-002010-39 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Avascular Necrosis of the Femoral Head
Keywords: avascular necrosis of femoral head; cell therapy; Mesenchymal stem cells
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultured autologous Mesenchymal Cells (Experimental): Cultured Mesenchymal Cells from bone marrow isolation, expanded under GMP protocol in associated facilities and introduced at the end of the appropriate forage up to the femoral head under fluoroscopic control.
  20x106 cells per cc in a single administration of 7cc
  Interventions: Biological: Cultured autologous Mesenchymal Cells

INTERVENTIONS:
Biological: Cultured autologous Mesenchymal Cells — Cultured Mesenchymal Cells from bone marrow isolation, expanded under GMP protocol in associated facilities and introduced at the end of the appropriate forage up to the femoral head under fluoroscopic control.

SUMMARY:
The purpose is to assess the safety and feasibility of cellular therapy derived from bone marrow, to help bone healing in patients with avascular necrosis of the hip.

DETAILED DESCRIPTION:
To assess the safety and feasibility of an in situ single injection of a high dose of autologous bone marrow-derived, in vitro expanded Mesenchymal stem cells, and its contribution to the resolution of the early stages of avascular osteonecrosis of the femoral head.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 65, both sexes

* Early avascular necrosis of the fem oral head (MRI diagnosis): Ficat and Arlet 0, 1, or 2 (Steinberg stages 0, I, IIA, IIB, or IIC)
* Sym ptom atic osteonecrosis with less than 6 months of evolution
* Able to provide informed consent, and signed informed consent
* Medical health care coverage

Exclusion Criteria:

* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control.
* Participation in another therapeutic trial in the previous 3 m onths
* Stages 3 or m ore (Ficat and Arlet) or III or m ore (Steinberg) of severe fem oral head osteonecrosis,primarily based on diagnosis by im aging (X-Rays, MRI).
* Flattening or collapse of the fem oral head (Steinberg stage IV) or articular cartilage collapse at the time of core decompression surgery.
* Septic arthritis.
* Stress fracture.
* Non-osteonecrosis metabolic bone diseases (particularly Paget's disease of bone, osteogenesis imperfecta, primary hyperparathyroidism , fibrous dysplasia monostotic, polyostotic McCune-Albright syndrome] and osteopetrosis).
* Any active bisphosphonate treatment or any history of intravenous (IV) treatment.
* History of prior or concurrent diagnosis of HIV-, Hepatitis-B- or Hepatitis-C-infection
* Active hepatitis B or hepatitis C infection at the time of screening.
* Known allergies to products involved in the production process of MSC.
* History of neoplasia or current neoplasia in any organ.
* Corticoid or immunosuppressive therapy more than one week in the two months prior to study inclusion
* Patients who will require continuous, systemic, high dose corticosteroid therapy (more than 7.5 m g/day) within 6 months after surgery.
* Patients who are in active treatment for cancer or blood dyscrasia, or have received chemotherapy, radiotherapy or immunotherapy in the past 2 years.
* History of regular alcohol consumption exceeding 2 drinks/day within 6 months of screening and/or history of illicit drug use.
* Serum AST (SGO T)/ALT (SGPT) > 2.5 X (institutional standard range).
* MRI-incompatible internal devices (pacemakers, aneurysm clips, etc).
* Body mass index (BMI) of 40 kg/m ² or greater.
* Patients unable to tolerate general anesthesia defined as an American Society of Anesthesiologists (ASA) criteria of > 2.
* Insulin dependent diabetes
* Patients with poorly controlled diabetes mellitus (HbA1C > 8%), or with peripheral neuropathy, or known concomitant vascular problems.
* Patients receiving treatment with hematopoietic growth factors or anti-vasculogenesis or antiangiogenesis treatment.
* Traumatic osteonecrosis.
* Adult in the care of a guardian (Subject legally protected)
* Im possibility to meet at the appointments for the clinical follow up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Complication rate | 12 months
  Includes early local complication rate plus global complication rate, as the percentage of patients with local or general complications at 52 weeks.

SECONDARY OUTCOMES:
complication rate | 6,12,24,104 weeks
  Local and general complication rate
Progression of disease to the next stage | 12 months
Amount of necrotic bone in the femoral head in MRI | 12 weeks and 52 weeks
Pain (VAS) | 6,12,24,52,104 weeks
serum levels of bone turnover markers | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gomez-Barrena, Prof, Study Chair — Universidad Autonoma de Madrid, Hospital la Paz
Locations (6):
- France (2):
  - Department of Orthopaedic Surgery, Hôpital Henri Mondor, Créteil
  - Department of Orthopaedic Surgery, CHU Tours, Tours
- Germany (2):
  - University Children's Hospital, Tübingen
  - Department of Orthopaedic Trauma, University of Ulm, Ulm
- Istituto Ortopedico Rizzoli, Bologna, Italy
- Servicio de Cirugía Ortopédica y Traumatología "A", Hospital La Paz, Madrid, Spain

REFERENCES:
- [Result] Gomez-Barrena E, Padilla-Eguiluz NG, Rosset P, Hernigou P, Baldini N, Ciapetti G, Gonzalo-Daganzo RM, Avendano-Sola C, Rouard H, Giordano R, Dominici M, Schrezenmeier H, Layrolle P, On Behalf Of The Reborne Consortium. Osteonecrosis of the Femoral Head Safely Healed with Autologous, Expanded, Bone Marrow-Derived Mesenchymal Stromal Cells in a Multicentric Trial with Minimum 5 Years Follow-Up. J Clin Med. 2021 Feb 1;10(3):508. doi: 10.3390/jcm10030508. PMID 33535589